CLINICAL TRIAL: NCT01163643
Title: A Randomized, Double-Masked, Parallel-Group, Vehicle Controlled, Multicenter, Exploratory Study Assessing the Safety and Efficacy of BOL-303242-X Ophthalmic Suspension in Dry Eye Syndrome
Brief Title: Study to Assess the Safety and Efficacy of BOL-303242-X Ophthalmic Suspension in Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 637
Record Dates: First submitted 2010-07-09; First posted 2010-07-16 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 0.3% BOL-303242-X ophthalmic suspension (Experimental): 0.3% BOL-303242-X ophthalmic suspension
  Interventions: Drug: 0.3% BOL-303242-X ophthalmic suspension
- 2% BOL-303242-X ophthalmic suspension (Experimental): 2% BOL-303242-X ophthalmic suspension
  Interventions: Drug: 2% BOL-303242-X ophthalmic suspension
- Vehicle (Placebo Comparator): Vehicle twice daily (BID)
  Interventions: Drug: Placebo Comparator: Vehicle
- 1% BOL-303242-X ophthalmic suspension (Experimental): 1% BOL-303242-X ophthalmic suspension
  Interventions: Drug: 1% BOL-303242-X ophthalmic suspension
- 2% BOL-303242-X ophthalmic suspension in the morning (Experimental): 2% BOL-303242-X ophthalmic suspension in the morning (AM) and vehicle in the afternoon (PM)
  Interventions: Drug: 2% BOL-303242-X ophthalmic suspension AM
- 2% BOL-303242-X ophthalmic suspension PM (Experimental): Vehicle in the AM and 2% BOL-303242-X ophthalmic suspension in the PM.
  Interventions: Drug: 2% BOL-303242-X ophthalmic suspension PM

INTERVENTIONS:
Drug: 0.3% BOL-303242-X ophthalmic suspension — 0.3% BOL-303242-X ophthalmic suspension BID for 12 weeks.
  Arms: 0.3% BOL-303242-X ophthalmic suspension
Drug: 2% BOL-303242-X ophthalmic suspension — 2% BOL-303242-X ophthalmic suspension BID for 12 weeks.
  Arms: 2% BOL-303242-X ophthalmic suspension
Drug: Placebo Comparator: Vehicle — Placebo Comparator: Vehicle BID for 12 weeks.
  Arms: Vehicle
Drug: 1% BOL-303242-X ophthalmic suspension — 1% BOL-303242-X ophthalmic suspension BID for 12 weeks.
  Arms: 1% BOL-303242-X ophthalmic suspension
Drug: 2% BOL-303242-X ophthalmic suspension AM — 2% BOL-303242-X ophthalmic suspension once daily (QD) AM and vehicle QD in PM for 12 weeks.
  Arms: 2% BOL-303242-X ophthalmic suspension in the morning
Drug: 2% BOL-303242-X ophthalmic suspension PM — Vehicle QD AM and 2% BOL-303242-X ophthalmic suspension QD in PM for 12 weeks.
  Arms: 2% BOL-303242-X ophthalmic suspension PM

SUMMARY:
The objective of this study is to identify the concentration and daily dosing frequency of BOL-303242-X ophthalmic suspension in treating dry eye syndrome over a 12 week dosing period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a diagnosis of dry eye disease.
* Intraocular pressure (IOP) ≤28 mmHg with no IOP lowering medications.
* Subjects who are willing and able to refrain from using contact lenses during the study.

Exclusion Criteria:

* Subjects with known hypersensitivity or contraindication to any component of the study medication.
* Subjects who are expected to require concurrent treatment with ophthalmic medications (prescription or over the counter).
* Subjects who are expected to require treatment with corticosteroids during the study.
* Subjects who have used topical or systemic isotretinoin, cyclosporine, or retinoid therapies within 30 days prior to the screening visit.
* Subjects who have undergone any type of ocular surgery within three months prior to screening.
* Lacrimal punctal occlusion (plugs or cautery) within 2 months of Screening Visit.
* Subjects with a history or presence of chronic generalized systemic or ocular disease that the Investigator feels might increase the risk to the subject or confound the result of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tuyen Ong, MD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2% BOL-303242-X Ophthalmic Suspension | 2% BOL-303242-X Ophthalmic Suspension in the Morning | 2% BOL-303242-X Ophthalmic Suspension PM | 1% BOL-303242-X Ophthalmic Suspension | 0.3% BOL-303242-X Ophthalmic Suspension | Vehicle
Started | 68 | 37 | 35 | 74 | 69 | 73
Completed | 62 | 35 | 33 | 69 | 61 | 66
Not Completed | 6 | 2 | 2 | 5 | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% BOL-303242-X Ophthalmic Suspension | 2% BOL-303242-X Ophthalmic Suspension in the Morning | 2% BOL-303242-X Ophthalmic Suspension PM | 1% BOL-303242-X Ophthalmic Suspension | 0.3% BOL-303242-X Ophthalmic Suspension | Vehicle | Total
Number analyzed (Participants) | 68 | 37 | 35 | 74 | 69 | 73 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (17.79) | 50.6 (16.99) | 51.8 (18.10) | 46.3 (17.64) | 46.5 (15.91) | 49.5 (17.56) | 48.4 (17.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 26 | 24 | 49 | 48 | 50 | 242
  Male | 23 | 11 | 11 | 25 | 21 | 23 | 114

OUTCOME MEASURES:

1. Primary Outcome: Mean Corneal Staining Score
Description: Total corneal staining score was calculated by adding the individual grades from 5 regions of the corneal surface (1: Central; 2: Superior; 3: Temporal; 4: Nasal; 5: Inferior). Grade 0 = none and Grade 3 = severe. The minimum total score possible was 0 and the maximum total score possible was 15. Higher scores indicated worse outcome.
Time Frame: 12 weeks
Population: Randomized participants with Week 12 results were included, with no imputation of missing data at Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2% BOL-303242-X Ophthalmic Suspension | 2% BOL-303242-X Ophthalmic Suspension in the Morning | 2% BOL-303242-X Ophthalmic Suspension PM | 1% BOL-303242-X Ophthalmic Suspension | 0.3% BOL-303242-X Ophthalmic Suspension | Vehicle
Number analyzed (Participants) | 64 | 35 | 33 | 71 | 64 | 67
score on a scale | 4.0 (3.19) | 3.9 (3.87) | 3.9 (3.66) | 4.4 (3.53) | 4.1 (3.03) | 3.7 (3.33)

2. Primary Outcome: Mean Worst Visual Analog Scale(VAS) Dry Eye Symptom
Description: Each symptom (ocular discomfort, dryness, grittiness, and stinging) was assessed to the nearest millimeter on a 0 - 10 cm Visual Analog Scale (VAS) by the subject. The worst VAS dry eye symptom was utilized in the analysis. The minimum for the worst symptom was 0 and the maximum for the worst symptom was 10.
Time Frame: 12 weeks
Population: Randomized participants with Week 12 results were included, with no imputation of missing data at Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2% BOL-303242-X Ophthalmic Suspension | 2% BOL-303242-X Ophthalmic Suspension in the Morning | 2% BOL-303242-X Ophthalmic Suspension PM | 1% BOL-303242-X Ophthalmic Suspension | 0.3% BOL-303242-X Ophthalmic Suspension | Vehicle
Number analyzed (Participants) | 64 | 34 | 33 | 71 | 65 | 67
score on a scale | 2.256 (2.3172) | 2.954 (2.4688) | 2.290 (2.4885) | 2.407 (2.6070) | 2.535 (2.5565) | 2.026 (2.1849)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The safety population included participants who received at least 1 dose of study drug. Participants confirmed to have never took a dose of study drug were excluded from safety analyses. Of the randomized participants, there was one 2% BOL-303242-X Ophthalmic Suspension participant, one 2% BOL-303242-X Ophthalmic Suspension PM participant, one 1% BOL-303242-X Ophthalmic Suspension participant, and 2 Vehicle participants who did not take at least one dose of study drug.
Arm/Group | 2% BOL-303242-X Ophthalmic Suspension | 2% BOL-303242-X Ophthalmic Suspension in the Morning | 2% BOL-303242-X Ophthalmic Suspension PM | 1% BOL-303242-X Ophthalmic Suspension | 0.3% BOL-303242-X Ophthalmic Suspension | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/37 | 0/34 | 0/73 | 0/69 | 0/71
Other Adverse Events (participants affected / at risk) | 1/67 | 2/37 | 1/34 | 2/73 | 3/69 | 5/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2% BOL-303242-X Ophthalmic Suspension (N=67) | 2% BOL-303242-X Ophthalmic Suspension in the Morning (N=37) | 2% BOL-303242-X Ophthalmic Suspension PM (N=34) | 1% BOL-303242-X Ophthalmic Suspension (N=73) | 0.3% BOL-303242-X Ophthalmic Suspension (N=69) | Vehicle (N=71)
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 1 | 2 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.